CLINICAL TRIAL: NCT02336659
Title: Influence of Gut Hormones on Food Intake After Roux-en-Y Gastric Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Maria Saur Svane, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MSV-14
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Severe Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — exendin (9-39); Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Saline (Placebo Comparator): Mixed meal test and ad libitum meal test duing infusion of saline
  Interventions: Other: Placebo
- Exendin 9-39 (Experimental): Mixed meal test and ad libitum meal test duing infusion of exendin 9-39, 900 pmol/kg/min
  Interventions: Drug: exendin 9-39
- DPP-4 Inhibition (Experimental): Mixed meal test and ad libitum meal test during intake of sitagliptin 100 mg * 2
  Interventions: Drug: sitagliptin
- Exendin 9-39 / DPP 4-Inhibition (Experimental): Mixed meal test and ad libitum meal test duing infusion of exendin 9-39, 900 pmol/kg/min and intake of sitagliptin 100 mg * 2
  Interventions: Drug: exendin 9-39; Drug: sitagliptin

INTERVENTIONS:
Drug: exendin 9-39 — Exendin 9-39 is a specific GLP-1 receptor antagonist
  Other Names: GLP-1 antagonist
  Arms: Exendin 9-39; Exendin 9-39 / DPP 4-Inhibition
Drug: sitagliptin — DPP-4 Inhibition
  Other Names: Januvia
  Arms: DPP-4 Inhibition; Exendin 9-39 / DPP 4-Inhibition
Other: Placebo — Saline
  Arms: Saline

SUMMARY:
The aim of this study is to examine the effect of GLP-1 and other gut-secreted hormones (glucagon, GIP, grelin and PYY) on food-intake, appetite and glucose metabolism after Roux-en-Y gastric bypass surgery.

DETAILED DESCRIPTION:
To do this the effect of combined GLP-1 receptor blockade by Exendin 9-39 and DPP-4-inhibition will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated RYGB performed 3-12 month proir to the study. Fasting plasma glucose <7.0 mM and HbA1c < 48 mmol/mol 3 month after RYGB.

Exclusion Criteria:

* Fasting plasma glucose >7.0 mM and HbA1c > 48 mmol/mol 3 month after RYGB. Hemoglobin <6.5mM. Previous anaphylaxis when treated with Januvia or Byetta. Allergy for sitagliptin. Dysregulated hypothyroidism. Use of antithyroid treatment. Late diabetic complications as retinopathy, renal insuffiency, neuropathy or previous pancreatitis. Bad compliance.
* Complications to RYGB: Documented reactive hypoglycaemia, severe dumping (with vomiting, diarrhea or severe abdominal pain after food intake).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-04; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Ad libitum food intake (changes in food intake) | 3-12 month after RYGB
  Evaluated by changes in food intake between the placebo day and the day with both administration of exendin 9-39 and DPP 4 Inhibitor

SECONDARY OUTCOMES:
Glucose metabolism (iAUC of glucose and c-pep after a meal) | 3-12 month after RYGB
  Evaluated by iAUC of glucose and c-pep after a meal
Gut-derived hormone profiles (iAUC of GLP-1, PYY, GIP and glucagon after a meal) | 3-12 month after RYGB
  Evaluated by iAUC of GLP-1, PYY, GIP and glucagon after a meal
Appetite measurement (VAS-scores) | 3-12 month after RYGB
  Evaluated by VAS-scores

CONTACTS AND LOCATIONS:
Overall Officials: Sten Madbad, MD, DMSc, Study Chair — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark